CLINICAL TRIAL: NCT07022080
Title: 68Ga-grazytracer PET/CT Study in Inflammatory Bowel Disease
Brief Title: Evaluating the Effectiveness of 68Ga-grazytracer PET/CT in Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252213
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases (IBD)
Keywords: PET/CT; 68Ga-grazytracer
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before-after study in the same patient (Experimental): About 69 patients with inflammatory bowel disease are planned to be included in this study. The screened subjects will undergo 68Ga-grazytracer PET/CT imaging before and at 2 weeks after drug therapy, and the investigators will collect clinical information from the patients, collect blood samples for granzyme B levels, and analyse the imaging results for data analysis.
  Interventions: Diagnostic Test: 68Ga-grazytracer PET/CT Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-grazytracer PET/CT Scan — The imaging agent 68Ga-grazytracer used in this project is synthesised in accordance with the standards for the production of radiopharmaceuticals with reference to the Chinese Pharmacopoeia (18F-FDG quality standard). pH value is between 5.0-8.0; radiochemical purity is not less than 95%, and the content of bacterial endotoxin per mL of solution is less than 15EU; the concentration of radioactivity is not less than 37MBq/mL; the solvent The residual amount of solvent complies with the regulations. Specification: 185~1850 MBq/ml Characteristics Colourless and transparent, no visible particles. Physical half-life: 68 minutes for 68Ga. Stable for 3 half-lives from the time of labelling. Method of administration: Intravenous. Dose: 0.05Ci/kg, followed by a 5 mL saline flush.

SUMMARY:
This is a single-centre, prospective, observational cohort study in which 69 patients with inflammatory bowel disease (IBD) were recruited to undergo 68Ga-grazytracer PET/CT imaging in patients with IBD to investigate the feasibility of early sensitive detection or prediction of the response to medication in patients with inflammatory bowel disease on 68Ga-grazytracer PET/CT and early prediction of the The feasibility of 68Ga-grazytracer PET/CT for early detection or prediction of response to drug therapy and early prediction of long-term prognosis in patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old; Clinical diagnosis of inflammatory bowel disease (active stage); Not having received treatment within 4 weeks prior to undergoing PET/CT examination; Received endoscopy within 7 days before and after PET/CT examination; Signing an informed consent form for PET/CT examination and volunteering to participate in this study.

Exclusion Criteria:

* No signed informed consent or unspecified diagnosis; Female subjects are pregnant or breastfeeding and male subjects are preparing for pregnancy; Those who are unfit to perform (concomitant severe and/or uncontrollable and/or unstable disease, developer allergy) or who are unable to complete imaging such as PET for specific reasons (needle-sickness, blood-sickness, claustrophobia); Colitis other than inflammatory bowel disease (infectious or ischaemic colitis); Patients who have undergone colon resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value | 1 day from injection of the tracer
  68Ga-grazytracer maximum standardised uptake value (SUVmax) in the subject's primary and/or lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, Shaanxi Province, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No